CLINICAL TRIAL: NCT06962007
Title: A Prospective, Randomized, Double-Blind Study of the Incidence, Severity, and Risk Factors of Clenching Induced by Sugammadex During Neuromuscular Blockade Reversal
Brief Title: Sugammadex-Induced Clenching During Neuromuscular Blockade Reversal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Cheol Lee,MD,PhD,, Professor, Wonkwang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Wonkwang UH17
Record Dates: First submitted 2025-04-27; First posted 2025-05-08 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Neuromuscular Blockade Reversal Agent; Perioperative Complications; Anesthesia, General; Sugammadex; Monitoring, Intraoperative; Masseter Muscle Spasm
Keywords: sugammadex; mouth clenching; neuromuscular blockade reversal
MeSH Terms: conditions — Trismus | interventions — Sugammadex; Population Groups; S 1 (combination); Epinephrine; Pyridostigmine Bromide

STUDY DESIGN:
Intervention Model Description: The study is not a safety/efficacy verification aimed at drug approval, but a mechanism/dose-related study to evaluate the dose-response and adverse event rate of already approved drugs.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sugammadex 1 mg/kg Group (S1) (Experimental): Participants receive 1 mg/kg of sugammadex intravenously for reversal of rocuronium-induced neuromuscular blockade.
  Interventions: Drug: Sugammadex 1 mg/kg Group
- Sugammadex 2 mg/kg Group (S2) (Experimental): Participants receive 2 mg/kg of sugammadex intravenously for reversal of rocuronium-induced neuromuscular blockade.
  Interventions: Drug: Sugammadex 2 mg/kg Group
- Sugammadex 4 mg/kg Group (S4) (Experimental): Participants receive 4 mg/kg of sugammadex intravenously for reversal of rocuronium-induced neuromuscular blockade.
  Interventions: Drug: Sugammadex 4 mg/kg Group
- Pyridostigmine/Glycopyrrolate Group (PG) (Active Comparator): Participants receive pyridostigmine 0.2 mg/kg and glycopyrrolate 0.01 mg/kg intravenously for reversal of rocuronium-induced neuromuscular blockade.
  Interventions: Drug: Pyridostigmine/Glycopyrrolate Group

INTERVENTIONS:
Drug: Sugammadex 1 mg/kg Group — Participants receive 1 mg/kg of sugammadex intravenously for reversal of rocuronium-induced neuromuscular blockade.
  Other Names: S1
  Arms: Sugammadex 1 mg/kg Group (S1)
Drug: Sugammadex 2 mg/kg Group — Participants receive 2 mg/kg of sugammadex intravenously for reversal of rocuronium-induced neuromuscular blockade.
  Other Names: S2
  Arms: Sugammadex 2 mg/kg Group (S2)
Drug: Sugammadex 4 mg/kg Group — Participants receive 4 mg/kg of sugammadex intravenously for reversal of rocuronium-induced neuromuscular blockade.
  Other Names: S4
  Arms: Sugammadex 4 mg/kg Group (S4)
Drug: Pyridostigmine/Glycopyrrolate Group — Participants receive pyridostigmine 0.2 mg/kg and glycopyrrolate 0.01 mg/kg intravenously for reversal of rocuronium-induced neuromuscular blockade.
  Other Names: PG
  Arms: Pyridostigmine/Glycopyrrolate Group (PG)

SUMMARY:
Study Objective:

This study aims to evaluate the incidence, severity, and risk factors of sugammadex-induced mouth clenching during neuromuscular blockade (NMB) reversal in adult surgical patients.

Study Design:

This prospective, randomized, double-blind, controlled clinical trial enrolls adult patients (ASA physical status I-II, aged 19-70 years) undergoing elective surgery under general anesthesia with rocuronium. Patients will be randomized into four groups to receive either sugammadex at doses of 1 mg/kg, 2 mg/kg, or 4 mg/kg, or a combination of pyridostigmine and glycopyrrolate.

Primary Outcome:

The primary outcome is the incidence of clenching within 10 minutes after NMB reversal, assessed by clinical observation, masseter EMG, and airway pressure changes, using a novel five-grade severity scale.

Secondary Outcomes:

Secondary outcomes include the severity of clenching, time to TOF ratio ≥0.9, BIS values at clenching onset, complications, and identification of risk factors such as dose, sex, BIS, age, BMI, and rocuronium dose.

Significance:

This study seeks to improve perioperative safety by identifying modifiable risk factors and informing dose adjustments or alternative reversal strategies to prevent sugammadex-induced clenching, particularly in high-risk populations.

DETAILED DESCRIPTION:
This prospective, randomized, double-blind clinical trial aims to investigate the incidence, risk factors, and clinical implications of sugammadex-induced clenching during neuromuscular blockade reversal under general anesthesia. Sugammadex, a selective relaxant binding agent, is widely used for the rapid reversal of rocuronium-induced neuromuscular blockade. However, reports of jaw clenching and masseter muscle contraction following sugammadex administration have raised safety concerns, particularly regarding airway management and patient discomfort during emergence from anesthesia.

A total of 240 adult patients (ASA physical status I-II, aged 19 to 70 years) scheduled for elective surgery under general anesthesia with rocuronium will be enrolled. Participants will be randomly assigned to one of four groups in a 1:1:1:1 ratio: sugammadex 1 mg/kg (S1), 2 mg/kg (S2), 4 mg/kg (S4), or pyridostigmine 0.2 mg/kg with glycopyrrolate 0.01 mg/kg (PG) as the control. Clenching events will be assessed within 10 minutes of drug administration using three criteria: visible jaw clenching, increased masseter electromyographic (EMG) activity (>50 μV for ≥2 seconds), and a rise in airway pressure (>5 cm H₂O). Severity will be graded using a novel five-level classification system.

Secondary outcomes include the severity and timing of clenching, time to train-of-four (TOF) ratio ≥0.9, bispectral index (BIS) value at the time of clenching onset, airway-related complications, and risk factor analysis based on dose, sex, BIS, age, BMI, and total rocuronium dose.

This study hypothesizes a dose-dependent increase in clenching with higher doses of sugammadex, potentially with a higher incidence in female patients and those with higher BIS values at reversal."

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants are adults aged 19-70 years, American Society of Anesthesiologists (ASA) physical status I-II, undergoing elective surgery under general anesthesia with rocuronium.

Exclusion Criteria:

* Exclusion criteria include neuromuscular disorders, renal impairment (creatinine clearance < 30 mL/min), history of clenching or dental disease, allergy to study drugs, or emergency surgery.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Incidence of Mouth Clenching After Neuromuscular Blockade Reversal | Within 10 minutes after administration of neuromuscular blockade reversal agent
  Clenching is defined as any of the following occurring within 10 minutes after administration of neuromuscular blockade reversal agents: (1) visible jaw clenching observed by the anesthesiologist, (2) masseter muscle electromyography (EMG) activity greater than 50 μV sustained for ≥2 seconds, or (3) airway pressure increase >5 cm H₂O.

SECONDARY OUTCOMES:
Severity of Mouth Clenching | Within 10 minutes after reversal agent administration
  Graded using a novel five-grade severity scale based on degree of jaw closure, EMG intensity, airway pressure, and need for intervention.
Time to Recovery of Train-of-Four (TOF) Ratio ≥0.9 | Up to 10 minutes after administration
  Measured using peripheral nerve stimulator; defined as time from reversal agent injection to TOF ratio ≥0.9.
Bispectral Index (BIS) at Clenching Onset | At time of clenching event, within 10 minutes post-reversal
  BIS value recorded at the time clenching is first detected.
Peak Airway Pressure | Within 10 minutes post-reversal
  Maximum airway pressure measured within 10 minutes after administration of reversal agent.
Incidence of Clenching-Related Complications | Within 10 minutes post-reversal
  Incidents such as bite injury, airway obstruction, or need for additional airway intervention during or after reversal.

CONTACTS AND LOCATIONS:
Overall Officials: Cheolhyeong Lee, MD, Principal Investigator — Wonkwang University Hospital
Locations (1):
- Wonkwang University hospital, Iksan, Jeonbuk-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in this article will be shared, including study protocol, statistical analysis plan, and analytic code.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 6 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal and agree to sign a data access agreement.

REFERENCES:
- [Background] Hristovska AM, Duch P, Allingstrup M, Afshari A. Efficacy and safety of sugammadex versus neostigmine in reversing neuromuscular blockade in adults. Cochrane Database Syst Rev. 2017 Aug 14;8(8):CD012763. doi: 10.1002/14651858.CD012763. PMID 28806470
- [Background] Naguib M. Sugammadex: another milestone in clinical neuromuscular pharmacology. Anesth Analg. 2007 Mar;104(3):575-81. doi: 10.1213/01.ane.0000244594.63318.fc. PMID 17312211
- [Background] Lee HY, Jung KT. Advantages and pitfalls of clinical application of sugammadex. Anesth Pain Med (Seoul). 2020 Jul 31;15(3):259-268. doi: 10.17085/apm.19099. PMID 33329823
- [Background] Lee S, Chung W. Sugammadex for our little ones: a brief narrative review. Anesth Pain Med (Seoul). 2024 Oct;19(4):269-279. doi: 10.17085/apm.24092. Epub 2024 Oct 31. PMID 39512049
- [Background] Tsur A, Kalansky A. Hypersensitivity associated with sugammadex administration: a systematic review. Anaesthesia. 2014 Nov;69(11):1251-7. doi: 10.1111/anae.12736. Epub 2014 May 22. PMID 24848211